CLINICAL TRIAL: NCT02719132
Title: A Multicentre Randomised Open-Label Crossover 2-Period 2 Treatment Clinical Trial to Evaluate Effect of Dapagliflozin 10 mg Once Daily on the Quality of Life in Patients With Type 2 Diabetes
Brief Title: Effect of DapagliFLOzin on Quality of Life in Patients With Type 2 Diabetes in a Real Clinical PrActice
Acronym: FLORA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1690C00043
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus type 2, dapagliflozin, quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 - therapy with dapagliflozin 10 mg once daily in combination with metformin ≤ 1,500 mg (daily dose) for 24 weeks (Treatment Regimen 1) followed by metformin monotherapy with dose titrated up to 2,500 mg/day for further 24 weeks (Treatment Regimen 2)
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Arm 2 (Active Comparator): Arm 2 - metformin monotherapy with dose titrated up to 2,500 mg/day for 24 weeks (Treatment Regimen 2) followed by therapy with dapagliflozin 10 mg once daily in combination with metformin ≤ 1,500 mg (daily dose) for further 24 weeks (Treatment Regimen 1)
  Interventions: Drug: Dapagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin, 10 mg
  Other Names: Forxiga
Drug: Metformin — Metformin, up to 2500 mg
  Other Names: Glucophage

SUMMARY:
This is a multicenter, randomised, open-label, crossover, 2-period comparative phase IV study.

The primary objective is to compare the effect of dapagliflozin 10 mg once daily in combination with metformin at a daily dose of ≤1,500 mg vs. metformin monotherapy with dose titrated up to 2,500 mg/day on the overall quality of life, obesity-specific quality of life and treatment satisfaction in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The study will comprise the following phases: Screening, Treatment Period 1 and Treatment Period 2.

After screening examinations and assessments, all patients enrolled will be randomly assigned in equal proportion (1:1) to either study arm:

Arm 1:

* Patients will take dapagliflozin 10 mg in combination with metformin ≤ 1,500 mg (daily dose) for 24 weeks during Treatment Period 1
* Patients will be on metformin monotherapy with dose titrated up to 2,500 mg/day for further 24 weeks during Treatment Period 2

Arm 2 (the same treatment phases in reverse order):

* Patients will be on metformin monotherapy with dose titrated up to 2,500 mg/day for 24 weeks during Treatment Period 1
* Patients will take dapagliflozin 10 mg in combination with metformin ≤ 1,500 mg (daily dose) for further 24 weeks during Treatment Period 2 Following the randomisation procedure, patients will receive investigational products at each visit as scheduled by Treatment Period 1. After the Randomisation Visit (Visit 2), the patient should attend the study centre for Visits 3, 4, and 5 (Day 28, Day 86, and Day 168, respectively) for efficacy and safety assessments. At Visit 5 (Day 168), the patient will receive investigational products as required by Treatment Period 2. Further Visits 6, 7 and 8 will be scheduled on Day 196, Day 252, Day 336, respectively.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients should fulfil ALL the criteria listed below:

1. A voluntary informed consent form for participation in the study signed by the patient prior to any study-specific procedures
2. Male and female patients of 18-74 years of age
3. Diagnosed type 2 diabetes
4. Therapy with metformin at a stable dose ≤1,500 mg/day for at least 8 weeks before enrolment
5. HbA1c >7.0% and ≤10% at the Screening Visit
6. C-peptide ≥1.0 ng/ml at the Screening Visit
7. Body mass index ≤45.0 kg/m² at the Screening Visit
8. For women of childbearing potential - use of reliable birth control methods
9. Ability to complete study-specific procedures
10. Ability to complete questionnaires

Exclusion Criteria:

1. Type 1 diabetes
2. Diabetic ketoacidosis at Screening
3. AST and/or ALT > 3 × upper limit of normal at Screening
4. Total serum bilirubin > 34.19 μmol/l at Screening
5. Decompensated diabetes mellitus (HbA1c >10% at Screening)
6. Patients with moderate to severe renal impairment (CrCl <60 ml/min or <60 ml/min/1.73 m2 at Screening) or terminal renal insufficiency
7. Severe concomitant diseases or severe cardiovascular, renal, hepatic, hematologic, endocrine, mental or rheumatic pathology
8. Malignancy within 5 years before enrolment
9. Acute (including viral and infectious) diseases within 1 month before the Screening Visit.
10. Development of severe acute diseases during the study which significantly affect the benefit/risk ratio for the subject or affecting study efficacy/safety assessment criteria
11. History of acute myocardial infarction or stroke within 6 months before the Screening Visit or during the study. Heart failure (NYHA III-IV)
12. Treatment with drugs affecting glucose homeostasis (e.g., systemic glucocorticosteroids) within 3 months before to the Screening Visit.
13. For women of childbearing potential - a positive pregnancy test or the patient is breast-feeding or planning pregnancy during the study
14. History of Hepatitis B and C or HIV
15. Individual hypersensitivity to any component of the investigational product (dapagliflozin)
16. Treatment with sodium-dependent glucose cotransporter inhibitors (SGLT2) has been administered within 3 months prior to enrolment or is planned during the study.
17. Loop diuretics have been administered for 3 months before the Screening Visit or are planned during the study.
18. Hereditary lactose intolerance, lactase deficiency and glucose-galactose malabsorption
19. The patient is unable to follow study procedures and attend the study centre for scheduled study visits or is going to relocate within the protocol-specific timelines
20. The patient is a subject of other studies within 3 months before enrolment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint including quality of life score | 48 weeks
  Change in the overall quality of life, obesity-specific quality of life and treatment satisfaction in the course of the therapy by the end of each 24-week treatment period compared to the quality of life, obesity-specific quality of life and treatment satisfaction at baseline.

SECONDARY OUTCOMES:
Change in HbA1c level | 48 weeks
  Change in HbA1c level will be assessed as mean change in the course of the treatment compared to baseline.
Change in body weight | 48 weeks
  Change in body weight will be assessed as mean change in body weight, mean percentage change in body weight and mean change in body mass index compared to baseline and as proportion of patients with body weight decreased by ≥5% during the treatment phase.
Change in waist circumference | 48 weeks
  Change in waist circumference will be assessed as mean change and mean percentage change in waist circumference during the treatment phase compared to baseline.
Change in fasting plasma glucose | 48 weeks
  Change in fasting plasma glucose will be assessed as mean change in fasting plasma glucose during the treatment phase compared to baseline.
Proportion of patients | 48 weeks
  Proportion of patients who achieved therapeutic glycaemic response (HbA1c ≤7%).

OTHER OUTCOMES:
ECG variables | 48 weeks
  ECG records including the following variables: heart rate (beats per minute), QT (msec), QTcB (msec), sinus heart rate (yes/no)
number of episodes of hypoglycaemia and ketoacidosis | 48 weeks
  number of episodes of hypoglycaemia and ketoacidosis
change in glomerular filtration rate | 48 weeks
  change in glomerular filtration rate compared to baseline at Screening
laboratory values changes | 48 weeks
  laboratory values (ALT, AST, total bilirubin, and creatinine)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Shestakova, Professor, Principal Investigator — Russian Federal Research Endocrinology center